CLINICAL TRIAL: NCT06780956
Title: Peri-implant Tissue Stability of Simplified vs Conventional Drilling Protocol Randomized Trial With 24-month Follow-up.
Brief Title: Simplified vs Conventional Drilling Protocol for Implant Placment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Artiom Lijnev, MSc, San Antonio Technologies - San Antonio Catholic University of Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE092002
Record Dates: First submitted 2024-10-24; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: MBL; Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional (Active Comparator): Conventional Drilling Protocol
  Interventions: Other: Conventional
- simplfied (Experimental): simplfied drilling protocol
  Interventions: Other: simplfied

INTERVENTIONS:
Other: Conventional — conventional drilling protocol using full sequence
  Arms: conventional
Other: simplfied — 3 burrs for implant placment
  Arms: simplfied

SUMMARY:
Despite the growing interest in these alternative drilling protocols, there is a lack of robust clinical evidence evaluating their long-term effects on MBL. The aim of the present study was therefore, to evaluate the effect of implant site preparation technique (conventional drilling versus simplfied) on change in the marginal bone level and insertion torque.

ELIGIBILITY:
Inclusion Criteria:

* Patients without any systemic pathologies that could be considered grounds for absolute contraindication.
* Adult patients who agreed to participate in the study and signed the informed consent form.
* Patients who smoked fewer than ten cigarettes per day.
* Patients who were not completely edentulous.
* Patients who were partially edentulous in the posterior maxillary or mandibular area and did not require the use of regenerative techniques.
* Patients with an area of healed, mature bone at least three months post-extraction.

Exclusion Criteria:

* Patients missing teeth in the esthetic zones 13-23 and 33-43 (second and fifth sextants).
* Patients who smoked more than ten cigarettes per day.
* Patients with a bleeding index greater than 30%.
* Patients with dental caries or periodontal disease.
* Pregnant or lactating women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss (MBL) | 24 month
  Is a non-infective remodeling process of variable entity occurring after implant placement.

CONTACTS AND LOCATIONS:
Locations (1):
- UCAM, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No